CLINICAL TRIAL: NCT06214169
Title: Effect of Addition of Cisatracurium to Lidocaine VS Plain Lidocaine for Intravenous Regional Anesthesia, a Comparative Study
Brief Title: Effect of Addition of Cisatracurium to Lidocaine VS Plain Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Muhammad Ilyas, Assistant Professor, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 446/23
Record Dates: First submitted 2023-12-26; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia
Keywords: Cisatracurium; Intravenous Regional Anesthesia; Lignocaine
MeSH Terms: interventions — cisatracurium; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain Lignocaine group (Other): Group of participants receiving only plain lignocaine for IVRA
  Interventions: Drug: Lignocaine
- Cisatracurium group (Other): Group of participants receiving plain lignocaine and cisatracurium combined for IVRA
  Interventions: Drug: Cisatracurium Besylate

INTERVENTIONS:
Drug: Cisatracurium Besylate — Addition of cisatracurium to plain lignocaine for IVRA.
  Arms: Cisatracurium group
Drug: Lignocaine — Plain Lignocaine for IVRA
  Arms: Plain Lignocaine group

SUMMARY:
The goal of this Randomized Control Trial is to compare the effects of addition of cisatracurium to lignocaine for IVRA Vs. Plain lignocaine in All ASA physical status I & II patients between 20 to 55 years of age, scheduled for elective hand surgery (carpal tunnel, trigger finger, tendon release, fracture reduction and tendon repair). The main question[s] it aims to answer are: • Does addition of Cisatracurium to plain lignocaine improve the overall quality of anesthesia? • Does use of cisatracurium lead to improved postop analgesia and decreased parenteral analgesic requirements? Participants will be Forty-four patients undergoing elective hand surgery during IVRA randomly assigned to two groups of 22 patients each. All demographic details (age, gender, body weight) will be noted, all will be briefed about visual analogue score (0 to 10) for pain. Group 1 (control group) will receive lidocaine 2% diluted with saline, group 2 (cisatracurium group) will receive cisatracurium plus lidocaine 2% diluted with saline. A standard technique would be employed for IVRA. The following parameters to be assessed: onset and offset of sensory and motor block, Intra-operative pain at 5, 10, 20, 30 minutes after tourniquet application by using visual analogue score (VAS), and postoperative pain using visual analogue score (VAS) measured at 5-minute,1, 2, 4, 8 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All ASA physical status I & II patients between 20 to 55 years of age, scheduled for elective hand surgery

Exclusion Criteria:

* Patients with Raynaud disease, sickle cell anemia, or a history of allergy to any drug to be used.
* Also, patients who had bleeding tendency, on anticoagulant or antiplatelet therapy, significant cardiovascular, peripheral vascular, or neurological disease.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Time to onset of Sensory blockade. | 1-5 min.
  Sensory block will be assessed by pinprick in the dermatomal sensory distribution and time noted for complete sensory blockade.
Time to onset of Motor Blockade | 2-7 min.
  Motor block will be assessed by asking the subject to flex and extend his/her wrist and fingers, every 30 seconds and time to be noted till inability to flex or extend the wrist and fingers is confirmed and time noted.
Intraoperative Pain Scoring | 5-45 min.
  The severity of intraoperative pain will be assessed using 10 point VAS (Visual Analogue Score) with 1 being no pain and 10 being the worst possible pain at 5, 10, 20, 30 minutes after tourniquet application.
Regression of sensory blockade | 2-10 min post deflation.
  Sensory blockade regression time (the time elapsed from tourniquet deflation to recovery of complete sensation in all dermatomes, determined by pinprick test) , will be noted.
Regression of motor blockade | 2-10 min post deflation
  Motor block regression time (the time elapsed from tourniquet deflation until regaining of flexion and extension of wrist and fingers) will be noted.
Postop Pain scoring | 5 minutes post deflaton till 8 hours post deflation.
  Postoperative pain will be assessed by VAS at 5 minutes after tourniquet deflation and at 1, 2, 4, 8 hours postoperatively.
Time to first analgesic request post operatively. | 1 hour - 8 hours post deflation.
  The first analgesic dose requirement time will also be noted (the time elapsed from tourniquet release until first request for analgesic medication postoperatively)
Side Effects | From onset of blockade to 8 hours post operatively.
  Incidence of side effects such as tinnitus, dizziness, convulsions, gastric discomfort, muscle weakness and bleeding tendency will be recorded intraoperatively as well as during recovery from blockade.

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Millitary Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prabhakar A, Lambert T, Kaye RJ, Gaignard SM, Ragusa J, Wheat S, Moll V, Cornett EM, Urman RD, Kaye AD. Adjuvants in clinical regional anesthesia practice: A comprehensive review. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):415-423. doi: 10.1016/j.bpa.2019.06.001. Epub 2019 Jul 2. PMID 31791560
- [Background] Esmaoglu A, Akin A, Mizrak A, Turk Y, Boyaci A. Addition of cisatracurium to lidocaine for intravenous regional anesthesia. J Clin Anesth. 2006 May;18(3):194-7. doi: 10.1016/j.jclinane.2005.08.003. PMID 16731321
- [Background] Farbood A, Khademi S, Tajvidi R, Hooshangi M, Salari S, Ghani M, Tahmasebi S, Jamali H. Comparison of Intravenous Regional Anesthesia with Single-Cuff Forearm Tourniquet and Hematoma Block and Traditional Method in Patients with Distal Radius Fractures; A Randomized Clinical Trial. Bull Emerg Trauma. 2020 Apr;8(2):77-82. doi: 10.30476/BEAT.2020.46446. PMID 32420391